CLINICAL TRIAL: NCT06919224
Title: Delivering Patient-Facing Evidence-Based Guidelines Through mHealth to Adults With Sickle Cell Disease (PF-Guide)
Brief Title: Delivering Patient-Facing Evidence-Based Guidelines Through mHealth to Adults With Sickle Cell Disease
Acronym: PF-Guide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Illinois at Chicago (Other); Washington University School of Medicine (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Robert Cronin, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL174590 (NIH)
Record Dates: First submitted 2024-04-22; First posted 2025-04-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth app + booklets (Active Comparator): A mHealth app that has patient facing guidelines and engaging content and a booklet with the guidelines that are made to be patient-facing.
  Interventions: Other: mHealth app + booklets
- Standard care (No Intervention): Group 1 will receive the control arm with standard care

INTERVENTIONS:
Other: mHealth app + booklets — A mHealth app that has patient facing guidelines and engaging content and a booklet with the guidelines that are made to be patient-facing.
  Arms: mHealth app + booklets

SUMMARY:
In a hybrid type I effectiveness-implementation trial, our three-center research teams aim to examine whether empowering adults with sickle cell disease (SCD) with patient-facing SCD-specific guidelines through an mHealth application with booklets will decrease acute healthcare utilization and be cost-effective over booklets with the guidelines alone. Our team, head will test our hypotheses with the following aims: Aim 1: evaluate the effectiveness of the patient-facing guidelines mHealth app + booklet intervention to decrease acute healthcare utilization (hospitalizations, emergency room visits, and day hospital visits) in adults with SCD over the standard care in a randomized controlled trial, Aim 2: evaluate the implementation outcomes of the mHealth app + booklet using the capability, opportunity, and motivation-behavior (COM-B) and reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) frameworks, and Aim 3: evaluate the cost-effectiveness of patient-facing mHealth app + booklets vs. standard care in adults with SCD. is hybrid effectiveness-implementation trial design, according to the COM-B and RE-AIM frameworks with a mixed-methods approach, will give valuable insights into the effects, facilitators, and barriers to the implementation that will influence the effects of the patient-facing guidelines intervention.

DETAILED DESCRIPTION:
The investigators propose a multi-center hybrid type I effectiveness-implementation trial to assess patient-facing evidence-based guidelines through a mHealth application plus (+) booklets in adults with sickle cell disease (SCD). Clinicians' care of SCD is informed by evidence-based guidelines, which can prevent morbidity and mortality. The National Heart, Lung, and Blood Institute (NHLBI) and the American Society of Hematology (ASH) published guidelines for evidence-based management of SCD for healthcare providers. However, patient, provider, or system barriers prohibit adequate reach within and across all three domains, leading to poor guideline adherence. Our prior work demonstrates 1) the patient's lack of knowledge of evidence-based guidelines, 2) the desire for guidelines to be patient-centered, accessible, and actionable in booklets and a mHealth app, 3) the development of patient-facing booklets with the guidelines and 4) the successful pilot of an engaging mHealth app with the guidelines that adults with SCD will use. Promising preliminary data from our multi-center feasibility randomized controlled trial support using a mHealth app + booklets with patient-facing guidelines for reducing acute healthcare utilization in adults with SCD. In the feasibility trial, the investigators screened 74 participants; 91% (67 of 74) agreed to be recruited and randomized to mHealth + booklet vs. booklets alone. A relative risk reduction of 44% occurred in acute healthcare utilization in the mHealth + booklet arm vs. the booklet alone arm. A total of 75% (50 of 67) of the participants agreed to be followed for six months to assess healthcare utilization and surveys of knowledge and patient-reported outcomes. Based on our preliminary trial results indicating a decrease of at least 44% in acute healthcare utilization (a decrease of 1.5 emergency room visits or hospital admissions per year) with mHealth + booklet, the investigators propose a three-center randomized controlled trial to test the following hypothesis: There will be a 44% relative risk reduction of acute healthcare utilization in adults with SCD (n=272), randomly allocated to mHealth app + booklets vs. standard care, defined as general guidance without patient-facing educational materials, for 12 months. The aims of this proposed study are Aim 1: evaluate the effectiveness of the patient-facing guidelines mHealth app + booklet intervention to decrease acute healthcare utilization (hospitalizations, emergency room visits, and day hospital visits) in adults with SCD over the standard care in a randomized controlled trial, Aim 2: evaluate the implementation outcomes of the mHealth app + booklet using the capability, opportunity, and motivation-behavior (COM-B) and reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) frameworks, and Aim 3: evaluate the cost-effectiveness of patient-facing mHealth app + booklets vs. standard care in adults with SCD. This hybrid effectiveness-implementation trial design, according to the COM-B and RE-AIM frameworks with a mixed-methods approach, will give valuable insights into the effects, facilitators, and barriers to the implementation that will influence the effects of the patient-facing guidelines intervention.

ELIGIBILITY:
Inclusion criteria for adults with SCD include

1. receiving care at the SCD clinic for the prior 12 months,
2. has a diagnosis of SCD (Hgb SS, SC, Sβ-thal),
3. able to speak and understand written English,
4. older than 18 years.

Inclusion criteria for the providers and staff members are

(1) to be involved in participants' clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Acute healthcare utilization | 12 month
  The investigators will measure a count of the # ER visits, # of hospitalizations, and # of day hospital visits (infusion center visits)

SECONDARY OUTCOMES:
Self-efficacy | 12 months
  sickle cell self-efficacy scale, as described in Edwards R, Telfair J, Cecil H, Lenoci J. Reliability and validity of a self-efficacy instrument specific to sickle cell disease. Behav Res Ther. 2000;38(9):951-63.
  Scale is 0-45, higher score is better Scale has no subscales and measures self-efficacy
SCD-specific knowledge | 12 months
  Knowledge about SCD guidelines. The knowledge part of the measure is a questionnaire that is multiple choice and asks questions about sickle cell disease with one correct answer and 3 incorrect answers. The investigators will sum up the number of correct answers to determine a score.
  This is not a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Cronin, MD, MS, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - University of Illinois at Chicago, Chicago, Illinois
  - Washington University St. Louis, St Louis, Missouri
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No